CLINICAL TRIAL: NCT01028261
Title: A Randomized, Double-Blind, Placebo-Controlled Multiple Dose Study, to Assess Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of ZGN-433 in Obese Volunteers
Brief Title: Safety, Tolerability and Pharmacokinetics of Multiple Doses of ZGN-433 in Obese Female Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zafgen, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZAF-001
Record Dates: First submitted 2009-12-07; First posted 2009-12-09 (Estimated); Last update posted 2012-01-11 (Estimated); Status verified 2012-01

CONDITIONS: Obesity
Keywords: Obese; Obesity; Overweight
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ZGN-433 (Experimental)
  Interventions: Drug: ZGN-433
- Normal Saline (Placebo Comparator)
  Interventions: Drug: ZGN-433

INTERVENTIONS:
Drug: ZGN-433 — Subjects will receive placebo or ZGN-433 twice weekly over 6 weeks treatment period for a total of 12 doses. A range of doses will be evaluated.
  Other Names: Beloranib hemioxalate

SUMMARY:
The purpose of this study is to assess whether multiple doses of ZGN-433 is safe and well tolerated in obese female subjects. The study will also provide information on how much ZGN-433 gets into the blood, how long does it stay in the body, and how it affects other biological markers.

DETAILED DESCRIPTION:
This protocol is designed to test the safety and preliminary efficacy of a drug called ZGN-433. It is to be tested for its ability to reduce weight in severely obese female subjects who are post menopausal or infertile.

ELIGIBILITY:
Inclusion Criteria:

* Obese, otherwise healthy females
* Post menopausal or infertile
* Weight ≥ 50 kg
* BMI ≥ 32 and ≤ 45 kg/m2

Exclusion Criteria:

* Use of weight loss agents in the past month
* History of eating disorder
* History of diabetes or other endocrine disorder
* History of gastric bypass
* Current smokers
* Unstable body weight during the past 3 months

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2009-12; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Measures of the safety and tolerability of ZGN-433 include documentation of adverse events and changes (compared to baseline) in vital signs, physical examination, heart rhythm, and laboratory tests. | Approximately 2 months

SECONDARY OUTCOMES:
Weight | Approximately 2 months

CONTACTS AND LOCATIONS:
Overall Officials: James E Vath, PhD, Study Director — Zafgen, Inc.
Locations (2):
- Australia (2):
  - Q-Pharm Clinics, Royal Brisbane and Women's Hospital, Brisbane, Queensland
  - Nucleus Network, Heidelberg, Victoria